CLINICAL TRIAL: NCT01897142
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo-controlled, Single Ascending Dose Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-05230907 In Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-05230907 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: B2341001; 2013-001387-36 (EudraCT Number)
Record Dates: First submitted 2013-06-24; First posted 2013-07-11 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — PF-05230907

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- PF-05230907 and Placebo Cohort 1 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907
- PF-05230907 and Placebo Cohort 2 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907
- PF-05230907 and Placebo Cohort 3 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907
- PF-05230907 and Placebo Cohort 4 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907
- PF-05230907 and Placebo Cohort 5 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907
- PF-05230907 and Placebo Cohort 6 (Experimental)
  Interventions: Biological: PF-05230907; Drug: Placebo for PF-05230907

INTERVENTIONS:
Biological: PF-05230907 — 0.1 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 1
Drug: Placebo for PF-05230907 — 0.1 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 1
Biological: PF-05230907 — 0.3 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 2
Drug: Placebo for PF-05230907 — 0.3 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 2
Biological: PF-05230907 — 1 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 3
Drug: Placebo for PF-05230907 — 1 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 3
Biological: PF-05230907 — 2 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 4
Drug: Placebo for PF-05230907 — 2 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 4
Biological: PF-05230907 — 3 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 5
Drug: Placebo for PF-05230907 — 3 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 5
Biological: PF-05230907 — 5 micrograms per kilogram of PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 6
Drug: Placebo for PF-05230907 — 5 micrograms per kilogram of placebo for PF-05230907, IV bolus, single dose
  Arms: PF-05230907 and Placebo Cohort 6

SUMMARY:
The purpose of this study is to determine what the study drug does to the body, what the body does to the study drug, and if the study drug is safe and well tolerated when given to adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects.
* Healthy non-child bearing female subjects.
* 18 to 35 years of age.

Exclusion Criteria:

* Heart disease.
* Clotting disorders.
* Use of nicotine products.
* Diabetes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting treatment related adverse events | Through Day 43
Incidence, severity and causal relationship of treatment emergent adverse events, treatment emergent serious adverse events, and withdrawals due to treatment emergent adverse events | Through Day 43
Incidence and magnitude of treatment emergent abnormal laboratory findings | Through Day 43
Change from baseline in vital sign measurements, ECG parameters, and physical examinations | Through Day 43

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Through 4 hour post dose Day 1
Maximum Observed Plasma Concentration (Cmax) | Through 4 hour post dose Day 1
Pharmacodynamic activity as measured by prothrombin time/internationalize normalized ration (PT/INR) | Through post dose Day3
Pharmacodynamic activity as measured by activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) | Through post dose Day3
Pharmacodynamic activity as measured by thrombin-antithrombin (TAT) complexes | Through post dose Day 2
Pharmacodynamic activity as measured by prothrombin fragments 1+2 (PF1+2) | Through post dose Day 2
Pharmacodynamic activity as measured by D-dimer | Through post dose Day 7
Pharmacodynamic activity as measured by protein C activity | Through post dose Day 2
Pharmacodynamic activity as measured by Factor V activity | Through post dose Day 3
Incidence of antibody immune response | Through post dose Day 43
Factor X activity | Through post dose Day 43

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2341001&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-05230907%20In%20Healthy%20Volunteers